CLINICAL TRIAL: NCT06565598
Title: Observation on the Efficacy of Single-layer Robot-assisted Transperitoneal Retroperitoneal Tubeless Radical Nephrectomy
Brief Title: Single-layer Robot-assisted Transperitoneal Retroperitoneal Tubeless Radical Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Xiushui (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSL2024005
Record Dates: First submitted 2024-08-15; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Nonfunctional Kidney; Renal Cancer
Keywords: Laparoscopic radical nephrectomy; Transperitoneal approach; Robotic surgery; Tubeless
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional robot-assisted transabdominal radical nephrectomy (No Intervention): Radical nephrectomy was performed through traditional robot-assisted transabdominal approach
- Traditional laparoscopic transabdominal radical nephrectomy (No Intervention): Traditional laparoscopic radical nephrectomy was performed
- Single-layer robot-assisted transperitoneal retroperitoneal tubeless radical nephrectomy (Experimental): Through a single-level surgical approach, surgical robot-assisted transperitoneal retroperitoneal radical nephrectomy was performed.
  Interventions: Procedure: Single-layer robot-assisted transperitoneal retroperitoneal tubeless radical nephrectomy

INTERVENTIONS:
Procedure: Single-layer robot-assisted transperitoneal retroperitoneal tubeless radical nephrectomy — Free through the single layer of the posterior abdominal cavity
  Other Names: Single layer approach
  Arms: Single-layer robot-assisted transperitoneal retroperitoneal tubeless radical nephrectomy

SUMMARY:
To investigate the effect of single-layer robot-assisted retroperitoneal approach for radical nephrectomy without tubularization

DETAILED DESCRIPTION:
In this study, a multi-center retrospective study was conducted to evaluate the clinical efficacy of single-layer robot-assisted peritoneal retroperitoneal radical nephrectomy in patients with nephrectomy, and to compare the safety and effectiveness of traditional robot-assisted peritoneal radical nephrectomy

ELIGIBILITY:
Inclusion Criteria:

* Patients with various causes requiring radical nephrectomy

Exclusion Criteria:

* patients who could not tolerate laparoscopic surgery for various reasons
* patients whose preoperative blood pressure and blood glucose were not controlled to normal
* patients with contralateral nonfunctioning kidney or solitary kidney
* Multiple organ surgery at the same time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | 24 months
  Blood loss during operation
postoperative time of getting out of bed | 24 months
  Time to get out of bed after surgery
postoperative hospital stay | 2-5 Days
  Length of hospital stay after surgery
Whether to convert to laparotomy or not | 24 months
  According to the surgical records in the medical records, whether the operation was converted to laparotomy was checked, and the data were recorded when collecting the data.
Operation time | 1-3 Hours
  Complete operative time
whether the tumor was completely removed | 24 months
  Observe whether the tumor is complete according to the naked eye after surgery，Record and record to the surgical record, record when collecting the receipt.

SECONDARY OUTCOMES:
Clavien-Dindo grading | 24 months
  Grade I : long-term pain, fever, continuous bleeding and exudate, transient intestinal obstruction ; grade II : need blood transfusion, pneumonia ; grade III : hematuria requiring cystoscopy ; level IV : renal insufficiency requiring hemodialysis, respiratory insufficiency requiring ICU treatment, and cardiac insufficiency requiring ICU care.

CONTACTS AND LOCATIONS:
Locations (1):
- First People 's Hospital of Xiushui, Jiujiang, China